CLINICAL TRIAL: NCT05944939
Title: "Post" Operative Assessment of Socket Healing With Placement of Concentrated Growth Factor in Impacted Mandibular Third Molar Socket
Brief Title: Assessment of Bone Density in Impacted Mandibular Third Molar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dow Dental
Record Dates: First submitted 2023-05-30; First posted 2023-07-14 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2022-10

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): After third molar extraction concentrated growth factor is palced in socket and closure with silk3.0 compare bone density with control group
  Interventions: Procedure: Surgical extraction of impacted third molar
- Control group (Experimental): After extraction closure with silk 3.0 compare bone density with cases
  Interventions: Procedure: Surgical extraction of impacted third molar

INTERVENTIONS:
Procedure: Surgical extraction of impacted third molar — After surgical extraction of mandibular impacted teeth concentrated growth factor placed in socket closure done with help of silk 3.0 suture

SUMMARY:
Preoperative radiograph will be taken to assess the type of impaction either mesioangular, horizontal, distoangular and check mouth opening. Two groups involve in my study. After taking consent from all patients in first group is control group open extraction of impacted mandibular third molar prepared concentrated growth factor placed in fresh socket closure done with silk 3.0. In second case group open extraction of impacted mandibular third molar is closure with silk 3.0 without placement of concentrated growth factor.

Bone density will assessed using cone beam computed tomography 3 month and 6month postoperatively.

DETAILED DESCRIPTION:
Total number of patients who will fulfill the inclusion criteria of the study will be included in the study from oral and maxillofacial surgery OPD of Dow University of health sciences dow dental college campus. Preoperative radiograph will be taken to assess the type of impaction either mesioangular, horizontal, distoangular and check mouth opening. Two groups involve in my study. After taking consent from all patients in first group is control group open extraction of impacted mandibular third molar prepared concentrated growth factor placed in fresh socket closure done with silk 3.0. In second case group open extraction of impacted mandibular third molar is closure with silk 3.0 without placement of concentrated growth factor.

CONCENTRATED GROWTH FACTOR PREPARATION:

Concentrated growth factor is prepared by using patients own venous blood 10ml drawn from patients radial forearm which placed in without anticoagulant solutions in a sterile vacuette tubes. Centrifuged 30 sec acceleration, 2 mint -2700rmp, 4mint 2400rmp, 4 mints -2700rmp,3 mints -3000rmp, 30 sec deceleration and stop.

Concentrated growth factor contain rich growth factor taken from tube with help of tweezer with cutting two phases with scissors where the center and bottom layers connected. When concentrated growth factor is separated a quantity of growth factors is present at interface between concentrated growth factor and erythrocyte layer. concentrated growth factor glue is mould and squeezed the liquid element, to obtain a concentrated growth factor membrane and that membrane will be stored in normal saline for future.

In second case group. After open extraction of impacted mandibular third molar fresh socket closure will be performed with silk 3.0. Same Postoperative instruction and medication will be given to all patients. Bone density will assessed using cone beam computed tomography 3 month and 6month postoperatively. Comparision between mesioangular with mesioangular, distoangular with distoangular, horizontal with horizontal , vertical with vertical.(11)The mean gray level histogram values of the cone beam computed tomography at extraction socket will be obtained through digora software , gray scale is a digital photograpy , computer generated imagery and colorimetry . For each defect a regions of intrest can be created for the defect region and one the surrounding bone using the freehand selection tool, the minimum safety distance from one pixel to any cortical structure has to be ensured,after creating region of intrest the analysis is performed and result is transferred directly to statical analysis sheet,(Geiger, Blem et al. 2016) The difference in mean grey level values at study and control sites were tabulated and compared bone density. The purpose of using mandibular third molar because third molar is most commonly impacted teeth and routinly extracted with number of complications being reported and overcome these complication we are using CGF in third molar socket

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age above 17 years
* Impacted mandibular third molar

Exclusion Criteria:

* Teeth require closed extraction
* Significant medical history ( e.g. uncontrolled diabetes mellitus )
* Patients with history of radiotherapy and chemotherapy
* Bleeding disorders
* Any pathology like tumor and cyst 6. Developmental disorder 7. Previously operated any surgery of jaw 8. cigarette smokers 9. Maxillary third molar

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2023-12-06 (Estimated)

PRIMARY OUTCOMES:
Measure of bone density with help of cone beam computerized tomography after 3 months and 6 months | 3 month and 6 month
  Cases compare with control with help of cone beam computerized tomography

CONTACTS AND LOCATIONS:
Overall Officials: D O W, Principal Investigator — Dow University of Health Sciences
Locations (2):
- Pakistan (2):
  - Dow Dental college Dow university of health sciences, Karachi, Sindh
  - Dow university of health sciences, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: Yes
Randmised control trial
Supporting Information: ICF
Time Frame: 6 month
Access Criteria: Bone density with cbct